CLINICAL TRIAL: NCT02131857
Title: The Effectiveness of a Systemic Mindfulness-based Intervention Program in a Cystic Fibrosis Clinic
Acronym: Mindfulness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, blau hannah, Director, Pulmonary Institute, Rabin Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RMC-0321-12-ctil
Record Dates: First submitted 2014-04-28; First posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Cystic Fibrosis
Keywords: Mindfulness; stress reduction
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Staff (Experimental): active interventional program based on Mindfulness training
  Interventions: Behavioral: active interventional program based on Mindfulness training
- Parents (Experimental): active interventional program based on Mindfulness training
  Interventions: Behavioral: active interventional program based on Mindfulness training
- Patients with CF (Experimental): active interventional program based on Mindfulness training
  Interventions: Behavioral: active interventional program based on Mindfulness training

INTERVENTIONS:
Behavioral: active interventional program based on Mindfulness training — active interventional program based on Mindfulness training

SUMMARY:
Hypothesis 1: Mindfulness is a feasible tool for use within a cystic fibrosis (CF) clinic

Hypothesis 2: Participants in the mindfulness intervention will show an increased level of quality of life post intervention with the Mindfulness course

Hypothesis 3. Levels of mindfulness:

Participants in the mindfulness intervention will report increased mindfulness levels post-program completion as compared to pre-program completion

Hypothesis 4. Levels of stress:

Participants in the mindfulness intervention will report lower levels of stress post-program completion as compared with pre-program commencement.

Hypothesis 5. Levels of residual depressive symptoms post-mindfulness intervention program: Residual symptoms of depression are a risk factor for relapse of depression. Post -program participants of mindfulness will purport fewer residual depressive symptoms compared with pre-program.

Hypothesis 6. CF is associated with severe neutrophilic inflammation of the airways. As mindfulness intervention has been shown to modulate immune system it may improve physical aspects of CF including markers of inflammation and markers of lung disease (lung function tests and rate of pulmonary exacerbations) and nutritional state.

DETAILED DESCRIPTION:
The study will be an active interventional program for approximately six months in duration. All participants will initially undergo an initial assessment interview. Personnel trained and certified in mindfulness-based stress reduction (MBSR) will run mindfulness-based groups in 6-8 weekly 1 1/2 hour sessions (the staff group will comprise of 6 sessions and the parents' and patients' groups will be 8 sessions long). Participants will learn and engage in various formal and informal meditation practices during experiential learning of skills, including concentration, mindfulness of thoughts, emotions, feelings and bodily sensations, decentering, and letting go. Each group will include both practical exercises and a psycho-educational component. Daily homework, an essential aspect of the course, will include meditation practices together with exercises designed to integrate application of awareness skills into daily life. On day 0, participants will complete a battery of questionnaires as well as tests of the physical status of CF disease. This battery will be repeated at 8 weeks, and again at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CF clinically and by sweat test and/ or genetic testing and/ or nasal potential difference
2. Treatment with one or more chronic medications or regimes;
3. Willingness by patient or parent to sign consent form;
4. Parents capable of complying with the program requirements including completing self-report questionnaires pre and post intervention completion.

Exclusion Criteria:

1. Having significant developmental delay or a mental health diagnosis of psychosis;
2. Transplant patients;
3. Participation in other interventional studies within 2 weeks of recruitment or during the study period -

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Score on the Mindful Attention Awareness Scale (MAAS) | 8 weeks
  The MAAS assesses individual differences in the frequency of mindful states over time and focuses on the presence or absence of attention to and awareness of what is occurring in the present. The MAAS includes a 15-item scale where respondents indicate how frequently they have the experience described in each statement using a 6-point Likert scale. Changes in MAAS-measured mindfulness pre-to post-intervention have been related to declines in mood disturbance and stress (reference #18).

SECONDARY OUTCOMES:
scores on the Cystic Fibrosis Questionnaire (CFQ-R) on 12 domains | 6 months
  The CFQ Is a disease-specific instrument designed to measure impact on overall health, daily life, perceived well-being and symptoms, developed specifically for use in patients with a diagnosis of cystic fibrosis. The measure consists of 12 subscales: Physical, Role, Vitality, Emotional State, Social/Marginalization, Body Image, Eating Disturbance, Treatment Burden, Perception of Health, Weight, Respiratory, and Digestion. Scores range from 0-100, with higher scores indicating better health-related quality of life (HRQOL). All subscales have been shown to have adequate internal consistency and test-retest reliability and have demonstrated good convergent and discriminant validity. (reference #17)
score on the Perceived Stress Scale (PSS) | 6 months
  Perceived Stress Scale (reference #19):
  The PSS measures the degree to which individuals perceive their daily life as being stressful during the last month with a 5-point Likert scale (0 = never and 4 = very often). Total scores can range from 0 to 40. Higher scores on the PSS represent higher levels of perceived stress.
Level of depression as assessed by the Beck Depression Inventory (BDI) | 6 months
  The BDI is a 21-item self - report measure of depressive symptoms. Each item presents one symptom at four levels of intensity scored from 0 to 3 yielding total scores ranging from 0 to 60, with 60 being the most extreme score of depression. The BDI has been found to be a reliable and valid measure of the severity of depressive symptoms in college students and adults (21) and in adolescents (22).
Pulmonary function as assessed by spirometry: forced expiratory volume in one second (FEV1), forced expiratory flow 25-75% (FEF25-75), and forced vital capacity (FVC) | 6 months
  The FEV1, FEF25-75 and FVC are assessed by spirometry techniques as done in the routine procedures in the Pulmonary clinic
CF related inflammation | 6 months
  levels of serum C-reactive protein (CRP), sputum neutrophil %,serum interleukin 8 (IL-8) and neutrophil elastase will be assessed by routine laboratory methods in the hospital laboratory
Rate of pulmonary exacerbations | 6 months
  the rate of pulmonary exacerbations will be assessed by the number of days on IV antibiotics as well as pulmonary exacerbations as defined by the FUCHS criteria
Score on the Mindful Attention Awareness Scale (MAAS) | 6 months
  The MAAS assesses individual differences in the frequency of mindful states over time and focuses on the presence or absence of attention to and awareness of what is occurring in the present. The MAAS includes a 15-item scale where respondents indicate how frequently they have the experience described in each statement using a 6-point Likert scale. Changes in MAAS-measured mindfulness pre-to post-intervention have been related to declines in mood disturbance and stress (reference #18).
scores on the Cystic Fibrosis Questionnaire (CFQ-R) on 12 domains | 8 weeks
  The CFQ Is a disease-specific instrument designed to measure impact on overall health, daily life, perceived well-being and symptoms, developed specifically for use in patients with a diagnosis of cystic fibrosis. The measure consists of 12 subscales: Physical, Role, Vitality, Emotional State, Social/Marginalization, Body Image, Eating Disturbance, Treatment Burden, Perception of Health, Weight, Respiratory, and Digestion. Scores range from 0-100, with higher scores indicating better health-related quality of life (HRQOL). All subscales have been shown to have adequate internal consistency and test-retest reliability and have demonstrated good convergent and discriminant validity. (reference #17)
score on the Perceived Stress Scale (PSS) | 8 weeks
  Perceived Stress Scale (reference #19):
  The PSS measures the degree to which individuals perceive their daily life as being stressful during the last month with a 5-point Likert scale (0 = never and 4 = very often). Total scores can range from 0 to 40. Higher scores on the PSS represent higher levels of perceived stress.
Level of depression as assessed by the Beck Depression Inventory (BDI) | 8 weeks
  The BDI is a 21-item self - report measure of depressive symptoms. Each item presents one symptom at four levels of intensity scored from 0 to 3 yielding total scores ranging from 0 to 60, with 60 being the most extreme score of depression. The BDI has been found to be a reliable and valid measure of the severity of depressive symptoms in college students and adults (21) and in adolescents (22).
Pulmonary function as assessed by spirometry: forced expiratory volume in one second (FEV1), forced expiratory flow 25-75% (FEF25-75), and forced vital capacity (FVC) | 8 weeks
  spirometry technique for measuring lung function
CF related inflammation | 8 weeks
  levels of serum C-reactive protein (CRP), sputum neutrophil %,serum interleukin 8 (IL-8) and neutrophil elastase will be assessed by routine laboratory methods in the hospital laboratory
Rate of pulmonary exacerbations | 8 weeks
  the rate of pulmonary exacerbations will be assessed by the number of days on IV antibiotics as well as pulmonary exacerbations as defined by the FUCHS criteria

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Blau, MBBS, Principal Investigator — Rabin Medical Center
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel